CLINICAL TRIAL: NCT00853008
Title: Treatment of High Risk Adult Acute Lymphoblastic Leukemia
Acronym: LAL-AR/2003
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-AR/2003
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; High-Risk (HR); Philadelphia Chromosome-Negative
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Daunorubicin; Prednisone; Mitoxantrone; Cytarabine; Dexamethasone; Methotrexate; Mercaptopurine; Teniposide; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vincristine — Vincristine (VCR): 1.5 mg/m2 (max 2 mg) IV d 1, 8, 15, 22 in induction VCR 2 mg, IV, d 1,8 in consolidation (cycle 1, 2)
Drug: Daunorubicin — Daunorubicin (DNR): 60 mg/m2 IV d 1, 8, 15, 22
Drug: Prednisone — Prednisone (PDN): 60 mg/m2/d IV or PO, d 1-28
Drug: Mitoxantrone — Mitoxantrone:12 mg/m2, IV d 15-17 in induction 12 mg/m2, IV,d 5 in cycle 2 consolidation
Drug: Cytosine Arabinoside — ARA-C 2,000 mg/m2/12h IV, d18,19 (4 doses) in induction
Drug: Dexamethasone — Dexamethasone 20 mg/m2,IV, d 1-5,10 mg/m2,IV, d 6 and 5 mg/m2,IV, d 7 in Consolidation (3 cycles)
Drug: Methotrexate (MTX) — Methotrexate (MTX)3 g/m2,IV, d1 (24h)in consolidation, cycles 1 and 2 MTX (15 mg/m2/wk, IM)in maintenance MTX 15 mg, IT
Drug: Cytarabine — Cytarabine 2g/m2/12h, IV d5 in cycle 1 consolidation Cytarabine 2g/m2/12h, IV d 1,2 in cycle 3 consolidation Cytarabine 30 mg, intrathecal
Drug: ASP — ASP 25,000 IU/m2, IV, d5 in consolidation (cycle 1, 2, 3)
Drug: Mercaptopurine — Mercaptopurine 100 mg/m2, PO, d 1-5 in consolidation
Drug: Teniposide — Teniposide 150 mg/m2, IV d 3,4 in consolidation cycle 3
Drug: Hydrocortisone — Hydrocortisone 20 mg, IT d 1, 28, 49, 77, 105, 175, 203, 231, 259,287, 311 intrathecal

SUMMARY:
Current therapeutic protocols for adult ALL consider MRD together with the baseline risk factors (age, WBC count, immunophenotype, cytogenetics) and speed in response to therapy for treatment decisions. On the other hand, the systematic use of allogeneic SCT for all adult patients (pts) with Ph- HR-ALL is still a matter of debate. The aim of the prospective study ALL-AR-03 from the Spanish PETHEMA Group was to evaluate the response to a differentiated therapy (chemotherapy or allogeneic SCT) according to early bone marrow blast clearance and MRD levels (assessed by cytofluorometry at the end of induction and consolidation therapy) in HR Ph- adult ALL patients.

DETAILED DESCRIPTION:
HR ALL included one or more of the following baseline parameters: age 30-60 yr, WBC count >25x109/L and 11q23 or MLL rearrangements. Induction therapy included vincristine, prednisone and daunorubicin for 4 weeks. In pts with slow cytologic response to therapy (≥10% blasts in bone marrow assessed on d14) intensified induction with high dose ARA-C and mitoxantrone was administered. Early consolidation therapy included 3 cycles with rotating cytotoxic drugs including high-dose methotrexate, high-dose ARA-C and high-dose asparaginase. Pts. with slow cytologic response on d14 or MRD level >0.05% after consolidation were assigned to allogeneic SCT (related or unrelated) and those with standard cytologic response on d14 and MRD level <0.05% after consolidation received 3 additional cycles of delayed consolidation (identical to those of early consolidation) followed by maintenance therapy up to 2yr in CR.

ELIGIBILITY:
Inclusion Criteria:

* High risk ALL adult patients (age> 15 years)no treated previously
* High-risk ALL:
* One or more of the following:

  * Age 30-60 yr.
  * WBC count >25x109/L
  * 11q23 or ALL1/AF4
* Very high-risk ALL:
* HR ALL and one or the following:

  * Slow cytologic response (>10% blasts in BM on d14 of induction therapy).
  * MRD>0.05% (by flow cytometry) at the end of consolidation

Exclusion Criteria:

* L3 ALL or B mature(sIg +) or t(8;14), t(2;8), t(8;22).
* ALL Ph (BCR/ABL) positive.
* Bifenotipics ALL as EGIL criteria.
* Indifferentiated ALL.
* Patients with cardiac pathology
* Patients with chronic liver disease in activity fase
* Pulmonary disease
* Renal insufficiency not due to ALL
* Neurological disorders not due to ALL
* PS (grades 3 and 4) not due to ALL.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the response to a differentiated therapy (chemotherapy or allogeneic SCT) according to early bone marrow blast clearance and MRD levels in HR Ph- adult ALL patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ribera Josep Mª, Dr, Study Chair — PETHEMA Foundation
Locations (38):
- Spain (38):
  - Hospital Juan Canalejo, A Coruña
  - Hospital General, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Clínica Teknon, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital Duran y Reynals, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital General, Castellon
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Josep Trueta, Girona
  - Hospital Universitario, Guadalajara
  - Hospital Xeral, Lugo
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico Universitario, Madrid
  - Hospital de Fuenlabrada, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Messeguer, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Llàtzer, Palma de Mallorca
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Parc Taulí, Sabadell
  - Hospital Clínico Universitario, Salamanca
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Xeral, Santiago
  - Hospital Virgen del Rocio, Seville
  - Hospital Joan XXIII, Tarragona
  - Hospital Mútua de Terrassa, Terrassa
  - Hospital Clínico Universitario, Valencia
  - Hospital Dr Pesset, Valencia
  - Hospital General, Valencia
  - Hospital La Fe, Valencia
  - Hospital Clínico, Valladolid
  - Hospital Virgen de la Concha, Zamora
  - Hospital Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Ribera JM, Oriol A, Morgades M, Montesinos P, Sarra J, Gonzalez-Campos J, Brunet S, Tormo M, Fernandez-Abellan P, Guardia R, Bernal MT, Esteve J, Barba P, Moreno MJ, Bermudez A, Cladera A, Escoda L, Garcia-Boyero R, Del Potro E, Bergua J, Amigo ML, Grande C, Rabunal MJ, Hernandez-Rivas JM, Feliu E. Treatment of high-risk Philadelphia chromosome-negative acute lymphoblastic leukemia in adolescents and adults according to early cytologic response and minimal residual disease after consolidation assessed by flow cytometry: final results of the PETHEMA ALL-AR-03 trial. J Clin Oncol. 2014 May 20;32(15):1595-604. doi: 10.1200/JCO.2013.52.2425. Epub 2014 Apr 21. PMID 24752047
- See also: Spanish Association of Hematology — http://aehh.org